CLINICAL TRIAL: NCT03672630
Title: Comparison of Two- Versus Three-antibiotic Therapy for Pulmonary Mycobacterium Avium Complex Disease
Acronym: MAC2v3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kevin Winthrop (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Jewish Health (Other); The University of Texas Health Science Center at Tyler (Other); University Health Network, Toronto (Other); New York University (Other); Medical University of South Carolina (Other); Mayo Clinic (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of California, San Diego (Other); Stanford University (Other); University of Kansas (Other); Vancouver Clinic (Unknown); University of California, San Francisco (Other); University of Washington (Other); Johns Hopkins University (Other); University of Miami (Other); Emory University (Other); University of Iowa (Other); University of North Carolina (Other); Temple University (Other); Loma Linda University (Other); Columbia University (Other); University of Wisconsin, Madison (Other); Northwell Health (Other); Kaiser Permanente (Other); James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Kevin Winthrop, Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18819; PCS-2017C2-7764 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Mycobacterium Avium Complex; Nontuberculous Mycobacterium Infection
Keywords: NTM; MAC; mycobacteria; nontuberculous mycobacteria; azithromycin; ethambutol; rifampin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Mycobacterium Infections, Nontuberculous; Mycobacterium Infections | interventions — Azithromycin; Ethambutol; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2-drug regimen (Active Comparator): This arm is a 3 time per week (TIW) treatment regimen that includes azithromycin 500 mg po + ethambutol 25 mg/kg Treatment changes are at the discretion of the treating physician and patient. Where possible, changes in dosing or frequency that allow the patient to continue taking the assigned drugs during the 12 months study period are preferred.
  Interventions: Drug: Azithromycin; Drug: Ethambutol
- 3-drug regimen (Active Comparator): This arm is a 3 time per week (TIW) treatment regimen that includes azithromycin 500 mg po + ethambutol 25 mg/kg + rifampin 600 mg Treatment changes are at the discretion of the treating physician and patient. Where possible, changes in dosing or frequency that allow the patient to continue taking the assigned drugs during the 12 months study period are preferred.
  Interventions: Drug: Azithromycin; Drug: Ethambutol; Drug: Rifampin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 500 MG Oral Tablet [ZITHROMAX]
  Other Names: Zithromax
Drug: Ethambutol — Ethambutol 25 mg/kg [MYAMBUTOL]
  Other Names: Myambutol
Drug: Rifampin — Rifampin 600 MG [RIFADIN]
  Other Names: Rifadin
  Arms: 3-drug regimen

SUMMARY:
NTM therapy consists of a multi-drug macrolide based regimen for 18-24 months. Treated patients frequently experience debilitating side effects, and many patients delay the start of antibiotic treatment due to these risks. Common side effects include nausea, diarrhea, and fatigue, and rare but serious toxicities include ocular toxicity, hearing loss, and hematologic toxicity. To date, most of the evidence underlying the current treatment recommendations has come from observational studies in which either a macrolide has been combined with rifampin and ethambutol, or in some cases combined with ethambutol alone. The proposed study will answer whether a third drug is necessary or whether taking two drugs can increase tolerability without a substantial loss of efficacy.

DETAILED DESCRIPTION:
Mycobacterium avium complex (MAC) are a subset of nontuberculous mycobacteria (NTM), environmental bacteria that can cause chronic, debilitating pulmonary disease, primarily affecting those over age 60. The goals of treatment are to improve symptoms, stop disease progression, and clear the infection. We propose to address a longstanding controversy in the therapy of pulmonary MAC disease, whether patients must take three antibiotics concomitantly, or if two are sufficient. The study is a multicenter randomized pragmatic clinical trial to compare azithromycin + ethambutol (2-drug therapy) vs. azithromycin + ethambutol + rifampin (3-drug therapy) for non-cavitary pulmonary MAC disease. All clinical outcomes will be considered standard of care and abstracted from clinical records. Therapy changes and adverse events will be recorded at routine visits. Health-related quality of life (HRQoL) and self-reported toxicity will be captured centrally in a web-based database, and CT scans will be read centrally. Co-primary outcomes are culture conversion and tolerability of treatment. The primary analysis for culture conversion will be conducted as a per-protocol non-inferiority analysis, and the primary analysis for tolerability will be conducted as an intention-to-treat superiority analysis.

ELIGIBILITY:
Inclusion Criteria:

* Culture positive pulmonary MAC meeting ATS/IDSA disease criteria
* Age over 18 years
* Ability to provide informed consent

Exclusion Criteria:

* Fibrocavitary disease
* Planned surgery for MAC disease
* Patients who have cumulatively taken 6 weeks or more of multi-drug antimicrobial treatment for MAC
* Patients who are currently taking or have taken multi-drug antimicrobial treatment for NTM within the prior 30 days
* Diagnosis of Cystic fibrosis
* Diagnosis of HIV
* History of solid organ or hematologic transplant
* Significant drug-drug interaction not clinically manageable in the opinion of the investigator
* Contraindication to any component of the study treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Acid-fast bacilli (AFB) culture negativity | 12 months post randomization
  Two consecutive negative AFB cultures by 12 months post randomization without reversion to positive
Therapy completion | 12 months post randomization
  The proportion of patients who complete 12 months of therapy on their assigned regimen with "satisfactory adherence". "Satisfactory adherence" is defined as taking 80% of their prescribed doses/not missing more than 75 days of treatment.

SECONDARY OUTCOMES:
QOL-B Respiratory Symptoms Score | 12 months post randomization
  Quality of Life-Bronchiectasis (QOL-B) with NTM module The QOL-B is a self-administered questionnaire that has been validated in patients with bronchiectasis. The questionnaire measures 8 separate domains: Physical Functioning, Role Functioning, Vitality, Emotional Functioning, Social Functioning, Treatment Burden, Health Perceptions, and Respiratory Symptoms.
NTM Symptoms Score | 12 months post randomization
  Quality of Life-Bronchiectasis (QOL-B) with NTM module The QOL-B is a self-administered questionnaire that has been validated in patients with bronchiectasis. The NTM module includes 4 additional domains: Eating Problems, Body Image, Digestive Symptoms, and NTM Symptoms. No total score is calculated.
PROMIS Fatigue 7a short form score | 12 months post randomization
  PROMIS Fatigue 7a short form score The PROMIS Fatigue item banks assess a range of self-reported symptoms over the past seven days, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. Each question has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. The lowest possible raw score (indicating the highest subjective level of fatigue) is 7; and the highest possible raw score (indicating the lowest subjective level of fatigue) is 35.
Fatigue AE proportion | Cumulative to 12 months
  Self-report, Moderate or worse
Gastrointestinal AE proportion | up to 12 months
  Self-report, Moderate or worse: Nausea, diarrhea, decreased appetite, OR abdominal pain
Liver AE proportion | up to 12 months
  Laboratory grade 2 or higher abnormality
Macrolide resistance | 12 months post randomization
  Susceptibility at last positive culture

CONTACTS AND LOCATIONS:
Overall Officials: Emily Henkle, PhD, MPH, Study Director — Oregon Health and Science University; Kevin L Winthrop, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (26):
- United States (25):
  - Loma Linda University Medical Center, Loma Linda, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - National Jewish Health, Denver, Colorado
  - University of Miami, Miami, Florida
  - Tampa VA Medical Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Louisina State University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Northwell Health, Manhasset, New York
  - New York University, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center, Tyler, Texas
  - University of Washington, Seattle, Washington
  - Vancouver Clinic, Vancouver, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A Full Data Package will be made available in a PCORI-designated repository. The Full Data Package includes the Analyzable Data Set, Full Protocol, metadata, data dictionary, full statistical analysis plan (including all amendments and all documentation for additional work processes), and analytic code from the PCORI-funded research project. The Analyzable Dataset includes a final cleaned and locked data set that contains all the data used in conducting the analyses reported in the PCORI Final Research Report and is de-identified in accordance with the HIPAA Privacy Rule (45 C.F.R. § 164.514(b)).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The dataset will be available after completion of the study and publication of results.
Access Criteria: Third party data requests will be reviewed by a committee, and approved requests will require a DUA.

REFERENCES:
- [Background] Henkle E, Hedberg K, Schafer S, Novosad S, Winthrop KL. Population-based Incidence of Pulmonary Nontuberculous Mycobacterial Disease in Oregon 2007 to 2012. Ann Am Thorac Soc. 2015 May;12(5):642-7. doi: 10.1513/AnnalsATS.201412-559OC. PMID 25692495
- [Background] Prevots DR, Shaw PA, Strickland D, Jackson LA, Raebel MA, Blosky MA, Montes de Oca R, Shea YR, Seitz AE, Holland SM, Olivier KN. Nontuberculous mycobacterial lung disease prevalence at four integrated health care delivery systems. Am J Respir Crit Care Med. 2010 Oct 1;182(7):970-6. doi: 10.1164/rccm.201002-0310OC. Epub 2010 Jun 10. PMID 20538958
- [Background] Winthrop KL, McNelley E, Kendall B, Marshall-Olson A, Morris C, Cassidy M, Saulson A, Hedberg K. Pulmonary nontuberculous mycobacterial disease prevalence and clinical features: an emerging public health disease. Am J Respir Crit Care Med. 2010 Oct 1;182(7):977-82. doi: 10.1164/rccm.201003-0503OC. Epub 2010 May 27. PMID 20508209
- [Background] Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. doi: 10.1164/rccm.200604-571ST. No abstract available. PMID 17277290
- [Background] Griffith DE, Brown-Elliott BA, Shepherd S, McLarty J, Griffith L, Wallace RJ Jr. Ethambutol ocular toxicity in treatment regimens for Mycobacterium avium complex lung disease. Am J Respir Crit Care Med. 2005 Jul 15;172(2):250-3. doi: 10.1164/rccm.200407-863OC. Epub 2005 Apr 28. PMID 15860751
- [Background] Lee H, Sohn YM, Ko JY, Lee SY, Jhun BW, Park HY, Jeon K, Kim DH, Kim SY, Choi JE, Moon IJ, Shin SJ, Park HJ, Koh WJ. Once-daily dosing of amikacin for treatment of Mycobacterium abscessus lung disease. Int J Tuberc Lung Dis. 2017 Jul 1;21(7):818-824. doi: 10.5588/ijtld.16.0791. PMID 28633708
- [Background] Peloquin CA, Berning SE, Nitta AT, Simone PM, Goble M, Huitt GA, Iseman MD, Cook JL, Curran-Everett D. Aminoglycoside toxicity: daily versus thrice-weekly dosing for treatment of mycobacterial diseases. Clin Infect Dis. 2004 Jun 1;38(11):1538-44. doi: 10.1086/420742. Epub 2004 May 5. PMID 15156439
- [Background] Winthrop KL, Ku JH, Marras TK, Griffith DE, Daley CL, Olivier KN, Aksamit TR, Varley CD, Mackey K, Prevots DR. The tolerability of linezolid in the treatment of nontuberculous mycobacterial disease. Eur Respir J. 2015 Apr;45(4):1177-9. doi: 10.1183/09031936.00169114. Epub 2015 Jan 22. No abstract available. PMID 25614169
- [Background] Miwa S, Shirai M, Toyoshima M, Shirai T, Yasuda K, Yokomura K, Yamada T, Masuda M, Inui N, Chida K, Suda T, Hayakawa H. Efficacy of clarithromycin and ethambutol for Mycobacterium avium complex pulmonary disease. A preliminary study. Ann Am Thorac Soc. 2014 Jan;11(1):23-9. doi: 10.1513/AnnalsATS.201308-266OC. PMID 24298907
- [Background] Griffith DE, Adjemian J, Brown-Elliott BA, Philley JV, Prevots DR, Gaston C, Olivier KN, Wallace RJ Jr. Semiquantitative Culture Analysis during Therapy for Mycobacterium avium Complex Lung Disease. Am J Respir Crit Care Med. 2015 Sep 15;192(6):754-60. doi: 10.1164/rccm.201503-0444OC. PMID 26068042
- [Background] Kobashi Y, Matsushima T, Oka M. A double-blind randomized study of aminoglycoside infusion with combined therapy for pulmonary Mycobacterium avium complex disease. Respir Med. 2007 Jan;101(1):130-8. doi: 10.1016/j.rmed.2006.04.002. Epub 2006 Jun 5. PMID 16750618
- [Background] Wallace RJ Jr, Brown-Elliott BA, McNulty S, Philley JV, Killingley J, Wilson RW, York DS, Shepherd S, Griffith DE. Macrolide/Azalide therapy for nodular/bronchiectatic mycobacterium avium complex lung disease. Chest. 2014 Aug;146(2):276-282. doi: 10.1378/chest.13-2538. PMID 24457542
- [Background] Adjemian J, Prevots DR, Gallagher J, Heap K, Gupta R, Griffith D. Lack of adherence to evidence-based treatment guidelines for nontuberculous mycobacterial lung disease. Ann Am Thorac Soc. 2014 Jan;11(1):9-16. doi: 10.1513/AnnalsATS.201304-085OC. PMID 24236749
- [Background] Koh WJ, Moon SM, Kim SY, Woo MA, Kim S, Jhun BW, Park HY, Jeon K, Huh HJ, Ki CS, Lee NY, Chung MJ, Lee KS, Shin SJ, Daley CL, Kim H, Kwon OJ. Outcomes of Mycobacterium avium complex lung disease based on clinical phenotype. Eur Respir J. 2017 Sep 27;50(3):1602503. doi: 10.1183/13993003.02503-2016. Print 2017 Sep. PMID 28954780
- [Background] Hernan MA, Robins JM. Per-Protocol Analyses of Pragmatic Trials. N Engl J Med. 2017 Oct 5;377(14):1391-1398. doi: 10.1056/NEJMsm1605385. No abstract available. PMID 28976864
- [Background] Murray EJ, Hernan MA. Adherence adjustment in the Coronary Drug Project: A call for better per-protocol effect estimates in randomized trials. Clin Trials. 2016 Aug;13(4):372-8. doi: 10.1177/1740774516634335. Epub 2016 Mar 7. PMID 26951361
- [Background] White IR, Royston P, Wood AM. Multiple imputation using chained equations: Issues and guidance for practice. Stat Med. 2011 Feb 20;30(4):377-99. doi: 10.1002/sim.4067. Epub 2010 Nov 30. PMID 21225900
- [Background] U.S. Food and Drug Administration. FDA Guideline: Evaluation of Gender Differences in Clinical Investigations - Information Sheet, July 22, 1993. Found at https://www.fda.gov/RegulatoryInformation/Guidances/ucm126552.htm. Last accessed 6/11/18.
- [Background] Henkle E, Novosad S, Siegel SA, Varley CD, Stadnik A, Winthrop KL. Northwest Biorepository of Nontuberculous Mycobacteria Patients- Baseline Characteristics. B25 NON-TUBERCULOUS MYCOBACTERIA: EPIDEMIOLOGY, DIAGNOSIS, AND TREATMENT: American Thoracic Society; 2016. p. A3018-A.
- [Derived] Henkle E, Quittner AL, Dieckmann NF, Franklin H, Brunton AE, Daley CL, Winthrop KL; MAC2v3 Investigators. Patient-Reported Symptom and Health-Related Quality-of-Life Validation and Responsiveness During the First 6 Months of Treatment for Mycobacterium avium Complex Pulmonary Disease. Chest. 2023 Jul;164(1):53-64. doi: 10.1016/j.chest.2023.02.015. Epub 2023 Feb 17. PMID 36803647